CLINICAL TRIAL: NCT00005154
Title: National Health and Nutrition Examination Survey IV (NHANES (IV)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1026
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2009-04-14 (Estimated); Status verified 2009-04

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension; Blood Disease; Lung Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hypertension; Hematologic Diseases; Lung Diseases

SUMMARY:
To supplement the fourth National Health and Nutrition Examination Survey protocol to include data on the common heart, vascular, lung, and blood diseases.

DETAILED DESCRIPTION:
BACKGROUND:

The first National Health and Nutrition Examination Survey (NHANES I) was conducted by the National Center for Health Statistics between 1971 and 1974. NHANES I was a clustered, multi-stage stratified probability sample of 23,808 individuals ranging in age from one to 74 years and drawn from the non-institutionalized civilian population of the United States. A random subsample of the 14,407 examined adults aged 25-74 were given supplemental questionnaires on cardiovascular and respiratory history.

In 1981, the National Institute on Aging and the NCHS began a follow-up of the original NHANES I cohort. In order to evaluate the usefulness of major epidemiological studies for predicting coronary heart disease in the United States population, the NHLBI added a Framingham model verification component to the follow-up. The risk factors (systolic blood pressure, serum cholesterol, and cigarette smoking) for death from coronary heart disease were compared using results from the seventh cohort examination of 1960-1964 as baseline in Framingham and the NHANES I examination of 1971-1974 as baseline for the NHANES I Epidemiologic Follow-up Study (NHEFS). The endpoint for each study was coronary heart disease death as coded from the death certificates. Results of the NHLBI portion of the follow-up demonstrated that the major risk factors for coronary heart disease mortality described in previous Framingham analyses were applicable to the United States white adult population.

In 1986, the total surviving cohort of NHANES I (approximately 12,500) were re-contacted in order to improve risk factor morbidity and mortality analyses. The NHLBI contributed to funding the NHANES III and currently contributes to funding NHANES IV. NHANES III incorporated features which distinguished it from earlier surveys in the series. The features included a longitudinal component, meaning that individuals were followed over time for vital statistics and re-examination, long-term biological specimen banking, and oversampling of Blacks and Hispanics. The component of additional questions and procedures provided information on the common heart, vascular, lung, and blood diseases, risk factors and elements of medical care. It also indicated how representative the NHLBI population-based epidemiologic studies were and to what extent the findings of these studies could be generalized to the United States population. The major NHLBI ongoing studies which were compared with NHANES III were the Coronary Heart Disease Risk Factor Development in Young Adults (CARDIA), Atherosclerosis Risk in Communities (ARIC), the Framingham Heart Study, and the Cardiovascular Health Study.

Field work for NHANES III began in September 1988. The first wave of data collection was completed from 1989 to 1991. The second wave of data collection was carried out from 1992 to 1994. ECG data were released to the public in 1998.

DESIGN NARRATIVE:

Beginning in 1981, NHLBI supplemented the NHANES examination protocol by including questions about history of heart, lung, and blood diseases, and their treatment. The examination also included the Rose questionnaires for angina, myocardial infarction and peripheral vascular disease, 12-lead electrocardiograms, questions about known and suspected risk factors including active and passive smoking, weight history, use of exogenous hormones, family history of heart, lung and blood diseases, and selected aspects of diet, psychosocial characteristics (depression, anxiety, social support, job control and demands, and anger experience and expression), and lifestyle. If feasible, 2-hour ECG Holter monitor records were obtained to identify and classify premature ventricular contractions and to detect episodes of ischemia. Pulmonary function tests were performed using standardized methods and strict quality assurance procedures and the American Thoracic Society-Division of Lung Diseases respiratory disease questionnaires were administered. Waist and hip girth measurements were obtained along with other anthropometric measures. Blood pressure determinations were made in the home as well as in the mobile examination center. Blood tests included lipids and lipoproteins, fibrinogen, hematocrit, white blood cell count, and differentials, fasting and post-challenge insulin and glucose concentrations, and nutritional biochemistries.

The NHLBI is currently supporting part of NHANES IV. NHANES IV is a study of a representative sample of approximately 30,000 of the non-institutionalized population of the United States, obtained through the use of a complex multi-stage sampling design using a combination of health questionnaire and physical exam. Each single year and any combination of consecutive years comprises a nationally representative sample which will facilitate linkage to other surveys that provide yearly estimates such as the Continuing Survey of Food Intake by Individuals and allow limited national estimates from NHANES IV each year. The NHLBI component obtains information on the prevalence and distribution of common heart, vascular, pulmonary and blood diseases. The core questionnaire is based on the Health Interview Survey (HIS), and provides information on disease, risk factors, and components of medical care. Through the use of a Mobile Exam Center (MEC), subjects throughout the country are administered a standardized physical exam to obtain data on blood pressure, venipuncture, spirometry, congestive heart failure (CHF), and ankle-arm blood pressures. Sub-populations of the U.S. of particular interest, including minorities and age groups of particular concern like the very young and the elderly, will be over-sampled. Specific objectives of NHANES IV include: ascertaining the prevalence of common heart, vascular, lung, and blood disease in a representative sample of the non-institutionalized population of the United States; estimating the frequency and distribution of known and suspected risk factors for these heart, vascular, lung, and blood disease; measuring associations between risk factors and diseases; ascertaining the frequency and distribution of medical, surgical, pharmacologic, and behavioral interventions used to prevent or treat heart, lung and blood diseases; measuring trends over time in heart, lung and blood diseases and risk factors; relating clinically manifest disease, risk factors, and components of medical care detected at the baseline examination to subsequent morbidity and mortality (detected by follow-up questionnaires and matching with the National Death Index); determining the extent to which findings in NHLBI populations-based epidemiological studies reflect national data and may be generalized to the U.S. population. A Central Lipid Laboratory will be established to: standardize for lipid measurements; accurately measure total cholesterol and HDL cholesterol for the entire NHANES IV sample population; and accurately measure triglycerides for the fasting NHANES IV population.

Phase I data from the first three years of the study were made available in June, 2002. Phase II data from NHANES IV became available in May, 2004.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1981-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bachorik — Johns Hopkins University

REFERENCES:
- [Background] Leaverton PE, Sorlie PD, Kleinman JC, Dannenberg AL, Ingster-Moore L, Kannel WB, Cornoni-Huntley JC. Representativeness of the Framingham risk model for coronary heart disease mortality: a comparison with a national cohort study. J Chronic Dis. 1987;40(8):775-84. doi: 10.1016/0021-9681(87)90129-9. PMID 3597679
- [Background] Gillum RF, Makuc DM. Serum albumin, coronary heart disease, and death. Am Heart J. 1992 Feb;123(2):507-13. doi: 10.1016/0002-8703(92)90667-k. PMID 1736588
- [Background] Gillum RF, Ingram DD, Makuc DM. White blood cell count, coronary heart disease, and death: the NHANES I Epidemiologic Follow-up Study. Am Heart J. 1993 Mar;125(3):855-63. doi: 10.1016/0002-8703(93)90181-8. PMID 8438715
- [Background] Linn S, Fulwood R, Carroll M, Brook JG, Johnson C, Kalsbeek WD, Rifkind BM. Serum total cholesterol: HDL cholesterol ratios in US white and black adults by selected demographic and socioeconomic variables (HANES II). Am J Public Health. 1991 Aug;81(8):1038-43. doi: 10.2105/ajph.81.8.1038. PMID 1853996
- [Background] Feibleib M, Rifkind B, Sempos C, et al: Methodological issues in the measurement of CVD risk factors: within-person variability in selected serum lipid measures - results from the Third National Health and Nutrition Examination Survey (NHANES III). Can J Cardiol, 9 (suppl D):87D-88D, 1993
- [Background] Johnson CL, Rifkind BM, Sempos CT, Carroll MD, Bachorik PS, Briefel RR, Gordon DJ, Burt VL, Brown CD, Lippel K, et al. Declining serum total cholesterol levels among US adults. The National Health and Nutrition Examination Surveys. JAMA. 1993 Jun 16;269(23):3002-8. PMID 8501842
- [Background] Winkleby MA, Kraemer HC, Ahn DK, Varady AN. Ethnic and socioeconomic differences in cardiovascular disease risk factors: findings for women from the Third National Health and Nutrition Examination Survey, 1988-1994. JAMA. 1998 Jul 22-29;280(4):356-62. doi: 10.1001/jama.280.4.356. PMID 9686553
- [Background] Burt VL, Cutler JA, Higgins M, Horan MJ, Labarthe D, Whelton P, Brown C, Roccella EJ. Trends in the prevalence, awareness, treatment, and control of hypertension in the adult US population. Data from the health examination surveys, 1960 to 1991. Hypertension. 1995 Jul;26(1):60-9. doi: 10.1161/01.hyp.26.1.60. PMID 7607734
- [Background] Andersen RE, Crespo CJ, Bartlett SJ, Cheskin LJ, Pratt M. Relationship of physical activity and television watching with body weight and level of fatness among children: results from the Third National Health and Nutrition Examination Survey. JAMA. 1998 Mar 25;279(12):938-42. doi: 10.1001/jama.279.12.938. PMID 9544768
- [Background] Gillum RF, Mussolino ME, Sempos CT. Baseline serum total cholesterol and coronary heart disease incidence in African-American women (the NHANES I epidemiologic follow-up study). National Health and Nutrition Examination Survey. Am J Cardiol. 1998 May 15;81(10):1246-9. doi: 10.1016/s0002-9149(98)00122-2. PMID 9604962
- [Background] Vargas CM, Ingram DD, Gillum RF. Incidence of hypertension and educational attainment: the NHANES I epidemiologic followup study. First National Health and Nutrition Examination Survey. Am J Epidemiol. 2000 Aug 1;152(3):272-8. doi: 10.1093/aje/152.3.272. PMID 10933274
- [Background] Fields LE, Burt VL, Cutler JA, Hughes J, Roccella EJ, Sorlie P. The burden of adult hypertension in the United States 1999 to 2000: a rising tide. Hypertension. 2004 Oct;44(4):398-404. doi: 10.1161/01.HYP.0000142248.54761.56. Epub 2004 Aug 23. PMID 15326093
- [Background] Carroll MD, Lacher DA, Sorlie PD, Cleeman JI, Gordon DJ, Wolz M, Grundy SM, Johnson CL. Trends in serum lipids and lipoproteins of adults, 1960-2002. JAMA. 2005 Oct 12;294(14):1773-81. doi: 10.1001/jama.294.14.1773. PMID 16219880
- [Derived] Xu Y, Yan Z, Liu L. Association between dietary intake of live microbes and chronic obstructive pulmonary disease: a cross-sectional study of NHANES 2007-2012. BMC Pulm Med. 2025 Jan 23;25(1):33. doi: 10.1186/s12890-024-03453-4. PMID 39849413
- [Derived] Lin Z, Zhu S, Cheng J, Lin Q, Lawrence WR, Zhang W, Huang Y, Chen Y, Gao Y. The mediating effect of engagement in physical activity over a 24-hour period on chronic disease and depression: Using compositional mediation model. J Affect Disord. 2022 Feb 15;299:264-272. doi: 10.1016/j.jad.2021.12.019. Epub 2021 Dec 11. PMID 34902506
- [Derived] Cameron NA, Petito LC, McCabe M, Allen NB, O'Brien MJ, Carnethon MR, Khan SS. Quantifying the Sex-Race/Ethnicity-Specific Burden of Obesity on Incident Diabetes Mellitus in the United States, 2001 to 2016: MESA and NHANES. J Am Heart Assoc. 2021 Feb 16;10(4):e018799. doi: 10.1161/JAHA.120.018799. Epub 2021 Feb 10. PMID 33563002